CLINICAL TRIAL: NCT00491283
Title: Comparison of Swab Types for Specimen Collection
Brief Title: QuickVue Influenza A+B Clinical Field Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quidel Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CS-0119-08(B)
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Swab Specimen Collection (QuickVue)

SUMMARY:
A comparative study of different swab types used for collection of specimens for rapid inluenza testing

ELIGIBILITY:
Inclusion Criteria:

Subjects must have:

* Fever (>38°C) (at time of visit or within the previous 48 hrs by history) and at least two of the following symptoms:

  * Chills/sweats
  * Cough
  * Dyspnea (labored, difficult breathing)
  * Fatigue
  * Headache
  * Myalgia (deep muscle aches)
  * Nasal congestion
  * Runny nose
  * Sore throat

Exclusion Criteria:

* Patients who are undergoing treatment with antivirals, now or within the last 7 days cannot be included in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | five months

SECONDARY OUTCOMES:
Sensitivity and Specificity | Positive and Negative Predictive Values

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Keller, MD, Principal Investigator — Sydney Airport medical Centre
Locations (1):
- Sydney Airport Medical Centre, Mascot, New South Wales, Australia